CLINICAL TRIAL: NCT01501474
Title: Utility of CholangioFlex and Fluorescent in Situ Hybridization in the Diagnosis of Malignant Biliary Strictures
Status: Terminated | Type: Observational
Why Stopped: No suitable case available and many techinical error
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, King Chulalongkorn Memorial Hospital, King Chulalongkorn Memorial Hospital
Other Study IDs: RP004
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Malignant Biliary Strictures
Keywords: Confocal; malignant biliary stricture; Sensitivity, specificity and accuracy of CholangioFlex in malignant biliary stricture diagnosis; sensitivity, specificity and accuracy of Fluorescent in situ Hybridization(FISH) in malignant biliary stricture diagnosis
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Brush cytology and FISH test
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CholangioFlex and Fluorescent in situ Hybridization(FISH)

SUMMARY:
Utility of CholangioFlex and Fluorescent in situ Hybridization in the Diagnosis of Malignant Biliary Strictures

Objectives

1. To assess the sensitivity, specificity and accuracy of CholangioFlex in malignant biliary stricture diagnosis
2. To assess the sensitivity, specificity and accuracy of Fluorescent in situ Hybridization(FISH) in malignant biliary stricture diagnosis

Study design One academic center, prospective, diagnostic study

Research Methodology Target population: Patients who are diagnosed malignant biliary stricture. Sample population: Patients who are diagnosed malignant biliary stricture in Chulalongkorn Hospital

DETAILED DESCRIPTION:
Utility of CholangioFlex and Fluorescent in situ Hybridization in the Diagnosis of Malignant Biliary Strictures

Objectives

1. To assess the sensitivity, specificity and accuracy of CholangioFlex in malignant biliary stricture diagnosis
2. To assess the sensitivity, specificity and accuracy of Fluorescent in situ Hybridization(FISH) in malignant biliary stricture diagnosis

Study design One academic center, prospective, diagnostic study

Research Methodology Target population: Patients who are diagnosed malignant biliary stricture. Sample population: Patients who are diagnosed malignant biliary stricture in Chulalongkorn Hospital

Inclusion Criteria

1. Age > 20 year-old
2. All patients who are diagnosed malignant biliary stricture by 3 months and undergo ERCP in Chulalongkorn Hospital.
3. All patients have to sign the consent form Exclusion Criteria

1.Cannot follow up for 1 year 2.Bleeding tendency including decompensated cirrhosis, chronic kidney disease and long-tem antiplatelets or anticoagulants 3.Pregnancy 4.History of fluorescein allergy

Timeline: From January 2012 to December 2013

Sample size Due to no study in Thai population before, investigator will perform pilot study in 50 malignant biliary stricture patients

Method

1. All patients had informed the consent.
2. Take the history, physical examination and then fill in the record form 3.5 ml of blood sampling for CA19-9 and 20 ml for further test by keeping in -20c temperature for 5 years

4.Set confocal endomicroscopy at the same session of ERCP 5.After successfully cannulation;

* 10% Fluorescein sodium 2.5 ml was injected intravenously.
* Confocal endomicroscopy (CholangioFlex) was performed at the suspected area. The video will record the images with Cellvizio program recorder.

  6.Brush cytology was performed 7.Record the duration and complication of the procedure 8.Send the tissues to one clinically-blinded GI pathologist for pathological diagnosis and FISH test 9.Compare the pathology and FISH report and endoscopic finding 10.Report the result According to Miami-criteria 2009, the Criteria for malignant biliary stricture from CholangioFlex are one of the followings;
  1. Thick branching bands (>20 microns)
  2. Dark clumps or glands (usually measuring > 60 microns)
  3. Bright and tortuous vessels

     Follow up
* The patients who are diagnosed malignant biliary obstruction will be treated as standard management
* The patients who are not diagnosed malignant biliary obstruction will be followed up every 3 months for 1 year
* The gold standard is pathology or clinical of malignancy including evidence of metastasis.

Statistical analysis Sensitivity, specificity, negative predictive value(NPV), positive predictive value(PPV) and accuracy by McNemar's test

Ethical considerations There is not a clearly evidence about the significant serious side effect of fluorescein injection. If the patients have side effects during the research, the procedure will be terminated and the patients will be in the responsibility of all investigators.

Expected benefit and application

1. Increase rate of malignant biliary stricture diagnosis by using CholangioFlex and/or FISH test
2. Decrease the mortality rate of malignant biliary stricture

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20 year-old
2. All patients who are diagnosed malignant biliary stricture by 3 months and undergo ERCP in Chulalongkorn Hospital.
3. All patients have to sign the consent form

Exclusion Criteria:

1. Cannot follow up for 1 year
2. Bleeding tendency including decompensated cirrhosis, chronic kidney disease and long-tem antiplatelets or anticoagulants
3. Pregnancy
4. History of fluorescein allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Due to no study in Thai population before, investigator will perform pilot study in 50 malignant biliary stricture patients
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Increasing the detection rate of malignant biliary stricture diagnosis by using CholangioFlex (Cofocal) and/or FISH test | up to 1 year
  If investigator can detect malignant biliary stricture more than present, the care giver can treat these patients properly. Consequently, the mortality rate of malignant biliary stricture will be decrease.

CONTACTS AND LOCATIONS:
Overall Officials: Rapat Pittayanon, MD, Principal Investigator — Chulalongkorn Hospital; Rungsun Rerknimitr, Professor, Study Director — Chulalongkorn Hospital
Locations (1):
- Rapat Pittayanon, Bangkok, Thailand

REFERENCES:
- See also: Related Info — http://www.medchulairb.com